CLINICAL TRIAL: NCT04630509
Title: Epidemiology and Outcomes of Pediatric Traumatic Cataract in Upper Egypt: A Tertiary Center Study
Brief Title: Epidemiology and Outcome of Pediatric Traumatic Cataract
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Mohamed M. A. Kedwany, Lecturer of Ophthalmology, Assiut University
Other Study IDs: Pediatric traumatic cataract
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Traumatic Cataract
Keywords: pediatric ocular trauma; Posterior chamber intraocular lens

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: traumatic cataract extraction — Irrigation/aspiration of traumatic cataract in children with posterior chamber intraocular lens implantation

SUMMARY:
this study aims to explore the demography of pediatric traumatic cataract in upper Egypt, and report outcomes and complications of traumatic cataract surgery in these children.

DETAILED DESCRIPTION:
Ocular trauma is one of the leading causes of acquired unilateral blindness in childhood.1,2 Apart from the permanent disability, ocular trauma has a profound impact on both patients and society at different levels, including, but not limited to, psychological trauma, cosmetic disfigurement, socioeconomic costs, and the need for specialized medical care and vocational rehabilitation.

Traumatic cataract is a common complication of pediatric eye injury. In developing countries, ocular trauma was responsible for up to 45% of childhood cataract. Vision loss induced by traumatic cataract is surgically manageable. However, the high risk of postoperative inflammation, posterior capsular opacification (PCO), amblyopia, and the associated ocular tissue damage may negatively impact visual outcome.

Several studies reported visual outcome of pediatric traumatic cataract in different populations. With the sacristy of studies on traumatic cataract in Egyptian children, we conducted this retrospective study to report the demographic features, visual outcome, and complications of pediatric traumatic cataract at Assiut University Hospital, the biggest tertiary referral center in Upper Egypt.

ELIGIBILITY:
Inclusion Criteria:

* All children who have undergone traumatic cataract surgery at Assiut university over 1 year period.

Exclusion Criteria:

* children with posterior segment injury.
* children who did not complete at least 6 months of postoperative follow-up.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children admitted for traumatic cataract surgery at Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Demographics | 6 months
  Age(in years), and gender (male or female) procedure, visual outcome, postoperative complications
Mechanism of injury | 6 months
  Blunt or penetrating eye injury
Visual outcome | 6 months
  Visual acuity according to Snellen chart and LogMAR

CONTACTS AND LOCATIONS:
Overall Officials: Salma Kedwany, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
to report the demographics and outcomes of pediatric traumatic cataract in upper Egypt

REFERENCES:
- [Derived] Kedwany SM, Saleh MGA, Tohamy D, Mostafa MM. Outcome of Pediatric Traumatic Cataract in Upper Egypt: A Tertiary Center Study. Clin Ophthalmol. 2021 Apr 16;15:1583-1589. doi: 10.2147/OPTH.S282080. eCollection 2021. PMID 33888974